CLINICAL TRIAL: NCT02937662
Title: Efficacy of Idarubicin, Cytarabine and Cyclophosphamide (IAC) Regimen in Relapsed/Refractory AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016006
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2019-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Cytarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IAC regimen (Experimental): Patients receive IAC regimen including idarubicin, cytarabine and cyclophosphamide.
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Drug: Cyclophosphamide
- Control Group (Active Comparator): Patients receive physician-directed regimens without cyclophosphamide including FLA±G regimen, AAG regimen, decitabine with AA regimen. Physicians can choose one of these regimens based on their experience and patients' condition.
  Interventions: Drug: Physician-Directed Regimens without Cyclophosphamide

INTERVENTIONS:
Drug: Idarubicin — Idarubicin at a dose of 10 mg/㎡/d on days 1-3.
  Arms: IAC regimen
Drug: Cytarabine — Cytarabine at a dose of 100mg/㎡/d on days 1-7.
  Other Names: Ara-c
  Arms: IAC regimen
Drug: Cyclophosphamide — Cyclophosphamide at a dose of 350mg/㎡/d on the second day and the fifth day.
  Other Names: CTX
  Arms: IAC regimen
Drug: Physician-Directed Regimens without Cyclophosphamide — Regimen without cyclophosphamide including FLA±G regimen, DA regimen, AAG regimen, decitabine with AA regimen.
  Arms: Control Group

SUMMARY:
In this multi-center, randomized, open-label, prospective clinical trial, a total of 60 relapsed/refractory AML patients will be randomized into 2 groups. In the experimental arm, patients receive IAC regimen. In the control arm, patients receive other physician-directed regimen. The primary end point is complete remission rate.

DETAILED DESCRIPTION:
In this multi-center, randomized, open-label, prospective clinical trial, a total of 60 relapsed/refractory AML patients will be randomized into 2 groups. Patients in the IAC arm receive the therapy consisting of idarubicin 10 mg/㎡/d on days 1-3, cytarabine 100mg/㎡/d on days 1-7 and cyclophosphamide at a dose of 350mg/㎡/d on the second day and the fifth day. In the control arm, patients received other physician-directed regimen including fludarabine, cytarabine with/without granulocyte stimulating factor(FLA±G) regimen,cytarabine plus daunorubicin(DA）regimen , decitabine,aclacinomycin and cytarabine(decitabine plus AA) regimen or AA regimen plus granulocyte stimulating factor. All the regimen in the control arm can not contain cyclophosphamide. The primary end point is complete remission. The second end points include overall survival, relapse-free survival and time to treatment failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age of less than 60 years old;
2. Patients that meet the diagnostic criteria(WHO 2008 criteria) of AML (except APL subtypes).
3. Patients with a confirmed pathologic diagnosis of AML which had relapsed or refractory.
4. Patients with ECOG score of ≤ 2;
5. Adult patients are willing to participate in the study and sign the informed consent by themselves or by their immediate family. Patients under 18 years old willing to participate should have their legal guardians sign the informed consent.

Exclusion Criteria:

1. Patients who had received reinduction therapy including cyclophosphamide are excluded. However, patients who had received regimens including cyclophosphamide before relapse are eligible.
2. Patients with other blood diseases(for example, haemophiliacs) are excluded.
3. Relapsed patients with only extramedullary leukemia;
4. After allogeneic hematopoietic stem cell transplantation;
5. With mutation of breakpoint cluster region-Abelson(BCR-ABL) fusion gene and in need of tyrosine kinase inhibitors therapy;
6. Acute panmyelosis with myelofibrosis and myeloid sarcoma patients;
7. Had other malignant tumor in need of treatment;
8. Had active cardiovascular disease;
9. Patients with other factors which were considered unsuitable to participate in the study by the investigators.

Ages: 0 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Complete Remission Rate | Within 6 weeks after induction therapy

SECONDARY OUTCOMES:
Overall Survival(OS) | Up to 3 years
  OS is defined as the time from the date of randomization until the date of death from any cause.
Relapse-Free Survival(RFS) | Up to 3 years
  RFS is defined as the time from the date of complete remission (CR) after entry in this trial until the date of documented relapse or death for subjects who achieve CR.
Time to Treatment Failure(TTF) | Up to 3 years
  TTF is defined as the time from the date of randomization until the date of death before response evaluation, not achieving CR or incomplete remission(CRi), or relapse/death after CR/CRi.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided